CLINICAL TRIAL: NCT03006211
Title: The Effects of Nitrogen Protoxide + Sevoflurane and Oxygen + Sevoflurane Anesthesia on Corneal Endothelial in Pediatric Patients
Brief Title: The Effects of Nitrogen Protoxide and Oxygen on Corneal Endothelial in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, M.D., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Asozkan-4
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Cornea; Anesthesia; Reaction
Keywords: nitrogen protoxide; oxygen; corneal endothelial; pediatric
MeSH Terms: conditions — Corneal Diseases | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- corneal endothal (Active Comparator): Evaluate the effects of nitrogen protoxide to corneal endothal and compare with oxygen.
  Interventions: Other: Nitrogen protoxide; Other: Oxygen
- Cell density (Active Comparator): Evaluate the effects of nitrogen protoxide to Cell density and compare with oxygen.
  Interventions: Other: Nitrogen protoxide; Other: Oxygen

INTERVENTIONS:
Other: Nitrogen protoxide
Other: Oxygen

SUMMARY:
To evaluate the mean changes in Endothelial Cell and Corneal pachymetry in eyes that operated under N2O + sevoflurane and O2 + sevoflurane general anesthesia.

DETAILED DESCRIPTION:
40 eyes of 40 patients who had extraocular surgery under general anesthesia will be included in this prospective study. Cell density, Cell variatio, Hexagonality rate and pachymetry specular microscopy results at before surgery and 1 week and 1 month after surgery will be analyzed. O2 (1 l/min) with 50% air and N2O (1 l/min) with 50% air will be applied to each group with flow rate 2 l/min totally, respectively. The duration of surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 40 eyes of 40 pediatric patients who had extraocular surgery under general anesthesia

Exclusion Criteria:

* None

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Change of corneal endothal number | after surgery at first day, 1th week and 1th month
  Nitrogen protoxide and oxygen may be change this number
Change of Cell density rate | after surgery at first day, 1th week and 1th month
  Nitrogen protoxide and oxygen may be change this rate
Change of Cell variation rate | at before surgery and 1 week and 1 month after surgery
  Nitrogen protoxide and oxygen may be change this rate
Change of Hexagonality rate | after surgery at first day, 1th week and 1th month
  Nitrogen protoxide and oxygen may be change this rate
Change of pachymetry specular microscopy results | after surgery at first day, 1th week and 1th month
  Nitrogen protoxide and oxygen may be change these results

IPD SHARING:
Plan to Share IPD: Undecided